CLINICAL TRIAL: NCT00297388
Title: A 52-wk Prospective, Randomized, Double-blind, Multicenter Study of Relapse Following Transition From Oral Antipsychotic Medication to 2 Different Doses (25 or 50 mg Every 2 Wks) of Risperidone Long-acting Microspheres (Risperdal� CONSTA�) in Adults With Schizophrenia or Schizoaffective Disorder
Brief Title: A Study of How Long it Takes a Patient to Relapse After Switching From an Oral Antipsychotic to One of Two Doses of Long-acting Risperidone Injections in Patients With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Janssen, LP (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002899
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; schizoaffective disorder; long-acting risperidone; intramuscular injection risperidone; risperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone, long-acting injectable

SUMMARY:
The purpose of this study is to assess the time for patients to relapse when switched from an oral antipsychotic to one of two doses of long-acting risperidone injection (shots). Risperidone has been used successfully to treat schizophrenia and schizoaffective disorder.

DETAILED DESCRIPTION:
Results from studies of older long-acting injectable antipsychotics (not risperidone) show that patients tend to relapse (which means start having symptoms again) when they are given low doses. However, increasing the dose may cause more side effects. This study will measure the time to relapse during a 52-week period in patients with schizophrenia or schizoaffective disorder who are switched from an oral antipsychotic (one taken by mouth) to one of two doses of long-acting risperidone injections (shots). The patients will be assigned to a dose of either 25 or 50 milligrams per injection every 2 weeks. Patients continue to take their usual oral antipsychotic medications up to 3 weeks following the first injection. After this 3-week period, they will receive the injectable risperidone only. Patients will be asked questions at each visit to help determine the effectiveness of the drug as assessed by the Clinical Global Impression Scale and the Positive and Negative Syndrome Scale. The safety of the drug will be based on patient signs and symptoms assessed according to the Extrapyramidal Symptom Rating Scale and self-reported treatment-emergent adverse events. Long-acting risperidone injection, 25 or 50 milligrams per injection, every 2 weeks for 52 weeks. Patients will continue to take their current oral antipsychotics for up to 3 weeks following the first injection of risperidone.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia or schizoaffective disorder
* stable with respect to disease symptoms and other medical conditions
* stable on any oral antipsychotic drug (except clozapine) for 4 weeks before the study
* patients identify a relative or acquaintance who can complete a questionnaire with additional information about the patient
* if female, using birth control.

Exclusion Criteria:

* Patient is not eligible if currently hospitalized, or was treated for an acute disease-related crisis within the past 4 weeks
* at risk to self or others
* use of injectable antipsychotic drugs or electroconvulsive therapy within past 6 months, or currently using carbamazepineor an oral antipsychotic drug in a dose that is higher than 8 milligrams per day in risperidone equivalents, of long-acting risperidone in an earlier study, of clozapine, or use of investigational drugs within 30 days, or of electroconvulsive therapy within past 6 months
* presence of liver or kidney damage
* history of neuroleptic malignant syndrome
* if pregnant or breast-feeding
* not using birth control
* abusing drugs or alcohol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Risperidone effectiveness is measured by time to relapse within the 52 week period.

SECONDARY OUTCOMES:
Effectiveness of the drug is assessed by the Clinical Global Impression Scale and Positive and Negative Syndrome Scale; safety as assessed by the Extrapyramidal Symptom Rating Scale and treatment-emergent adverse events during the 52 week period.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Simpson GM, Mahmoud RA, Lasser RA, Kujawa M, Bossie CA, Turkoz I, Rodriguez S, Gharabawi GM. A 1-year double-blind study of 2 doses of long-acting risperidone in stable patients with schizophrenia or schizoaffective disorder. J Clin Psychiatry. 2006 Aug;67(8):1194-203. doi: 10.4088/jcp.v67n0804. PMID 16965196
- See also: A 52-week, prospective, randomized, double-blind, multicenter study of relapse following transition from oral antipsychotic medication to two different doses of risperidone long-acting microspheres in adults with schizophrenia or schizoaffective disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=500&filename=CR002899_CSR.pdf